CLINICAL TRIAL: NCT01139528
Title: Conservative Treatment Versus Operative Treatment of Extra-articular Fractures in the Neck of the 5th Metacarpal Bone- A Prospective Randomized Trial
Brief Title: Conservative or Operative Treatment of Fractures in the Neck of the 5th Metacarpal Bone
Acronym: MC-studien
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: University Hospital, Akershus (Other); Asker & Baerum Hospital (Other)
Responsible Party: Principal Investigator, Ida Neergård Sletten, Consultant orthopaedic surgeon, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FASUUS 1529
Record Dates: First submitted 2010-05-18; First posted 2010-06-08 (Estimated); Last update posted 2015-04-24 (Estimated); Status verified 2015-04

CONDITIONS: Fractures of the Neck
Keywords: Fracture; 5th metacarpal bone; Bouquet pinning; Fractures of the neck of the 5th metacarpal bone
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Operative treatment (Active Comparator): Closed reduction of the fracture and osteosynthesis with 2-3 intramedullary K-wires (Bouquet method), cast treatment for 7-10 days followed by 5 weeks of buddy-strapping before removal of the K-pins
  Interventions: Procedure: Bouquet pinning of the 5th metacarpal bone
- Conservative treatment (No Intervention): No attempt of reduction of the fracture, 7-10 days of cast treatment followed by 5 weeks of buddy-strapping

INTERVENTIONS:
Procedure: Bouquet pinning of the 5th metacarpal bone — The fracture is reduced under general anesthesia and 2-3 K-pins are introduced in the medullar cavity to keep the fracture in the reduced position
  Arms: Operative treatment

SUMMARY:
A multi-site randomized controlled trial where patients are allocated to operative treatment or conservative treatment of fractures of the neck of the 5th metacarpal bone. The study goal is to identify which degree of angular displacement in the fracture that requires operative intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age with fractures of the neck of the 5th metacarpal bone

Exclusion Criteria:

* Less than 30 degrees of volar angulation in the fracture
* rotational deformity
* pseudoclawing
* intra-articular involvement
* ad latus displacement more than one half of a bone width
* concomitant fractures or soft tissue damage
* admittance more than 14 days after injury
* non-compliant patient (language, drugs, tourist)
* patient who refuses to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2010-05; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Quick-DASH | 6 weeks, 3 months, 1 year, 2 years
  Validated hand function score

SECONDARY OUTCOMES:
Patient satisfaction | 6 weeks, 3 months, 1 year, 2 years
  VAS scale
Pain | 1 week, 6 weeks, 3 months, 1 year, 2 years
  VAS scale
Eq-5d | 6 weeks, 3 months, 1 year, 2 years
  Validated quality of life score
Complications | 1 week, 6 weeks, 3 months, 1 year, 2 years
  All complications are noted
Sick-leave | 1 week, 6 weeks, 3 months (1 year, 2 years)
  Days of sick-leave off work
Range of motion in the joints in the 5th finger measured by hand therapist | 3 months, 1 year, 2 years
  total active motion 5th finger, totale passive motion 5th finger, active and passive extension and flexion in the 5th MCP-joint
Grip strength | 3 months, 1 year, 2 years
  Compared to the non-injured hand
Angular displacement in fracture measured in lateral x-ray, and shortening in fracture measured in AP view, of the 5th ray of the hand | 6 weeks, 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Lars Nordsletten, Prof. MD, PhD, Study Chair — University of Oslo
Locations (1):
- Oslo University Hospital, Oslo, Norway

REFERENCES:
- [Derived] Sletten IN, Nordsletten L, Hjorthaug GA, Hellund JC, Holme I, Kvernmo HD. Assessment of volar angulation and shortening in 5th metacarpal neck fractures: an inter- and intra-observer validity and reliability study. J Hand Surg Eur Vol. 2013 Jul;38(6):658-66. doi: 10.1177/1753193412461582. Epub 2012 Oct 11. PMID 23060463